CLINICAL TRIAL: NCT01503073
Title: Noninvasive Brain Stimulation for Stroke Improvement
Brief Title: Noninvasive Brain Stimulation for Stroke
Acronym: NIBSstroke
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professor, MD, PhD, University Hospital of Mont-Godinne
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B03920073136
Record Dates: First submitted 2011-12-23; First posted 2012-01-02 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real stimulation (Active Comparator): real NIBS
  Interventions: Device: tdcs (ELDITH, Neuroconn, Ilmenau, Germany)
- Sham stimulation (Sham Comparator): sham NIBS
  Interventions: Device: tdcs (ELDITH, Neuroconn, Ilmenau, Germany)

INTERVENTIONS:
Device: tdcs (ELDITH, Neuroconn, Ilmenau, Germany) — transcranial direct current stimulation

SUMMARY:
Noninvasive brain stimulations will be used in acute and chronic stroke patients to improve a variety of functions.

DETAILED DESCRIPTION:
Noninvasive brain stimulations (NIBS) will be used in acute and chronic stroke patients to improve a variety of functions such as motor functions, cognitive functions, ...

NIBS will be applied in a placebo-controlled, double-blind, randomised fashion. Behavioural data will be collected before and after NIBS, as well as brain functional imaging data.

ELIGIBILITY:
Inclusion Criteria:

* stroke with at least slight deficit

Exclusion Criteria:

* epilepsy
* contraindication to tDCS and/or to fMRI
* presence of metal in the head
* unability to understand / complete behavioural tasks
* chronic intake of alcohol or recreative drugs
* major health condition
* presence of pacemaker
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
change in function before/after tDCS | Before intervention, immediately after intervention, 10-20-30-40-50-60 min after intervention; long-term after intervention : 1-2-3-4 weeks, 2-3-4-5-6-7-8-9-10-11-12 months
  any brain function impaired by stroke

SECONDARY OUTCOMES:
change in neuroimaging and neurophysiological before/after tDCS | Before intervention, immediately after intervention, 10-20-30-40-50-60 min after intervention; long-term after intervention : 1-2-3-4 weeks, 2-3-4-5-6-7-8-9-10-11-12 months
  1. noninvasive neuroimaging : brain activity studied by means of fMRI
  2. noninvasive neurophysiological measure : TMS, EEG,evoked potentials, EMG

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, CHU Mont-Godinne, Yvoir, Namur, Belgium

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411
- [Derived] Lefebvre S, Thonnard JL, Laloux P, Peeters A, Jamart J, Vandermeeren Y. Single session of dual-tDCS transiently improves precision grip and dexterity of the paretic hand after stroke. Neurorehabil Neural Repair. 2014 Feb;28(2):100-10. doi: 10.1177/1545968313478485. Epub 2013 Mar 13. PMID 23486918